CLINICAL TRIAL: NCT02284659
Title: Effect of Functional Electrical Stimulation on Erectile Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Cristiane Carboni, Professor, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUHSPortoAlegre
Record Dates: First submitted 2014-10-31; First posted 2014-11-06 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FES-sham (Sham Comparator): Functional Electro Stimulation (FES-sham)
  Interventions: Device: FES- Sham
- Intervention (FES) (Active Comparator): functional electro stimulation
  Interventions: Device: Functional Electrical Stimulation (FES)

INTERVENTIONS:
Device: Functional Electrical Stimulation (FES) — FES (50Hz / 500us)
  Arms: Intervention (FES)
Device: FES- Sham
  Arms: FES-sham

SUMMARY:
Objective: The aim of this study is to evaluate the FES effect on erectile function in men with erectile dysfunction.

Expected Results: The hypothesis is that treatment with FES decrease erectile dysfunction.

DETAILED DESCRIPTION:
Introduction: Erectile dysfunction (ED) affects approximately 150 million men worldwide. The application of functional electrical stimulation (FES) has been used due to the high regenerative capacity of smooth muscle cells. This approach can be beneficial in the treatment of which usually has the ultimate causes cavernous smooth muscle degeneration.

Objective: The aim of this study is to evaluate the FES effect on erectile function in men with erectile dysfunction.

Methods: Randomized Clinical Trial will be selected in which 30 patients with erectile dysfunction. The men included will be randomized into two groups. The intervention group will conduct therapy with FES (50Hz / 500us) for 15 minutes with intensity below the motor threshold and the control group will use FES placebo. Two sessions will be held weekly for four weeks. Erectile function will be assessed using the validated questionnaire IIEF-5. The instrument will be completed by blinded researcher and the technique is randomized and the treatment done randomly.

Expected Results: The hypothesis is that treatment with FES decrease erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Male patient
* 40 to 65 years of age, with stable marital relationship (6 months)
* Diagnosis of erectile dysfunction (score of less than 22 IIEF5)
* Clinical history of ED for at least 6 months

Exclusion Criteria:

* A neurogenic (spinal cord injury, Parkinson's, MS, post prostatectomy)
* Hypogonadism (total testosterone <300 ng / dl)
* Patient reporting use of inhibitors or 5PDE FIC in the last 60 days
* Diagnosis of coronary artery disease and / or cerebrovascular disease
* Impossibility of understanding the goals, technical study and informed consent cognitive impairment

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-11; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Erectile function with International Index of Erectile Function-5 questionnaire | 2 times a week for 30 minutes